CLINICAL TRIAL: NCT00999063
Title: Prevalence of GERD in Patients With upperGITsymptoms in Thailand
Brief Title: Prevalence of Gastroesophageal Reflux Disease (GERD) in Patients With Upper Gastrointestinal Track (GIT) Symptoms in Thailand
Acronym: GerdQ
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sompob Paibulsirijit, MD, Vice President Medical& Regulatory Affairs department, AstraZeneca
Other Study IDs: NIS-GTH-NEX-2009/1
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Upper GIT Symptoms
Keywords: GerdQ

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a prospective , epidemiological, multi-centre, phase IV study, approximately 5,000 patients who suffer with upper gastrointestinal tract symptoms. Each patient will be assessed for GERD with GerdQ Thai Version.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Female or male aged at least 18 years
* Patient must be having symptoms suggestive of upper gastrointestinal tract symptoms such as heart burn/ regurgitation

Exclusion Criteria:

* Involvement in the planning and /or conduct of the study (applies to both AstraZeneca staff and /or staff at study site
* Participation in a clinical study(excluding non-interventional study or registry) during the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 4108 (Actual)
Dates: Start 2009-12; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Prevalence of gastroesophageal reflux disease (GERD) in patients presented with upper gastrointestinal tract symptoms

SECONDARY OUTCOMES:
Response to various treatments for patients who have been diagnosed of GERD

CONTACTS AND LOCATIONS:
Overall Officials: Somchai Leelasukolvong, Dr., Principal Investigator — Siriraj Hospital
Locations (25):
- Thailand (25):
  - Research Site, Bangkok Noi, Bangkok
  - Research Site, Muang, Bangkok
  - Research Site, Pathumwan, Bangkok
  - Research Site, Rajthevee, Bangkok
  - Research Site, Ratchthewi, Bangkok
  - Research Site, Maung, Changwat Khon Kaen
  - Research Site, Muang, Changwat Nonthaburi
  - Research Site, Klong Luang, Changwat Pathum Thani
  - Research Site, Maung, Changwat Ratchaburi
  - Research Site, Maung, Changwat Samut Sakhon
  - Research Site, Maung, Changwat Sukhothai
  - Research Site, Maung, Changwat Trang
  - Research Site, Muang, Changwat Udon Thani
  - Research Site, Maerim, Chiang Mai
  - Research Site, Maung, Chiang Mai
  - Research Site, Maung, Nakhon Sri Thammarat
  - Research Site, Maung, Nakhonratchasima
  - Research Site, Maung, Nakhonsawan
  - Research Site, Maung, Nakornpathom
  - Research Site, Maung, Phetchabun
  - Research Site, Maung, Phuket
  - Research Site, Maung, Roiet
  - Research Site, Maung, Ubonratchathani
  - Research Site, Varin Chamrap, Ubonratchathani
  - Research Site, Maung, Uttaradit